CLINICAL TRIAL: NCT00313508
Title: A Dose Ranging Trial of MART-1/gp100/Tyrosinase/NY-ESO-1 Peptide-Pulsed Dendritic Cells Matured Using Cytokines With Autologous Lymphocyte Infusion With or Without Escalating Doses of Fludarabine for Patients With Chemotherapy-naive Metastatic Melanoma
Brief Title: Dendritic Cell Vaccination During Lymphoid Reconstruction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13649; NCI-6241 (Other: NCI Protocol Number)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2012-12

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma; ciliary body and choroid melanoma, medium/large size; recurrent intraocular melanoma; metastatic intraocular melanoma; extraocular extension melanoma; iris melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Heart Rate; gp100 Melanoma Antigen; CTAG1B protein, human; MAGEA3 protein, human; Monophenol Monooxygenase; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Peptide-pulsed DC, ALI and Low Dose Fludarabine (Experimental): Fludarabine: 5 mg/m^2/day, Auto Lymphocyte Infusion, DC Infusion
  Interventions: Biological: Autologous Dendritic Cells (DC); Drug: Fludarabine; Biological: Autologous Lymphocyte Infusion (ALI)
- B: Peptide-pulsed DC, ALI and High Dose Fludarabine (Experimental): Fludarabine: 25 mg/m^2/day, Auto Lymphocyte Infusion, DC Infusion
  Interventions: Biological: Autologous Dendritic Cells (DC); Drug: Fludarabine; Biological: Autologous Lymphocyte Infusion (ALI)

INTERVENTIONS:
Biological: Autologous Dendritic Cells (DC) — Given intranodally
  Other Names: Autologous Dendritic Cells (DC) pulsed with tumor antigen class I peptides derived from MART-1 (26-35) (27L), gp100; (209-217 (210M), gp100 280-288 (288V), NY-ESO-1 157-165 (165V) and tyrosinase 207-215; as well as class II MART-1 (51-73), NY-ESO-1 (119-143), MAGE-3 (243-258) and tyrosinase; (450-462) peptides preceded by Autologous Lymphocyte Infusion (ALI) and one of two doses of; Fludarabine.
Drug: Fludarabine — Fludarabine will be administered intravenously (IV) over 30 minutes, daily for 5 consecutive days.
  Other Names: fludarabine phosphate; FLUDARA
Biological: Autologous Lymphocyte Infusion (ALI) — Infusion
  Other Names: ALI

SUMMARY:
This is a randomized, controlled, multicenter, dose-escalation study of fludarabine. Patients are randomized to 1 of 2 treatment arms.

The purpose of this study is to find out what side effects are caused in this study and whether Fludarabine with the dendritic cell vaccine (DC vaccine) can increase the ability of the immune system to recognize melanoma.

DETAILED DESCRIPTION:
This is a dose ranging study of intranodal administration of autologous dendritic cells (DC) pulsed with tumor antigen class I peptides derived from MART-1 (26-35) (27L), gp100 (209-217 (210M), gp100 280-288 (288V), NY-ESO-1 157-165 (165V) and tyrosinase 207-215 as well as class II MART-1 (51-73), NY-ESO-1 (119-143), MAGE-3 (243-258) and tyrosinase (450-462) peptides preceded by Autologous Lymphocyte Infusion (ALI) and one of two doses of Fludarabine. The nine or ten amino acid peptides representing HLA-A2 restricted T cell epitopes of MART-1, gp100, NY-ESO-1 and tyrosinase will be pulsed onto autologous dendritic cells produced by incubation of peripheral blood mononuclear cells obtained by apheresis with interleukin-4 (IL-4) and GM-CSF and pulsed with four helper peptides then matured with a cytokine cocktail including TNF-a, IL-6, IL-1b and PGE2. Melanoma antigen peptide-pulsed dendritic cells will be administered at a total dose of 10 million cells each for four intranodal injections to patients with chemotherapy-naïve metastatic melanoma.

DC matured with a cytokine cocktail and pulsed with class I and II peptides will be injected intranodally, weekly for two doses, then every two weeks for two doses, for a total of four injections to each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic melanoma with measurable disease after attempted curative surgical therapy and without prior chemotherapy; adjuvant interferon or isolated limb perfusion is allowed.
* Tumor tissue must be available for immunohistochemical analysis, and specimens will stained for MART-1/tyrosinase/NY-ESO-1 by immunohistochemical staining and will also be stained for HMB-45 by immunohistochemistry, and positivity for at least one will be an entry requirement.
* Patients must be HLA-A *0201 positive by a DNA polymerase chain reaction (PCR) analysis.
* Serum creatinine of 2.0 mg/dl or less, total bilirubin of 2.0 mg/dl or less, and alanine transaminase/aspartic transaminase (ALT/AST) of less than 3X institutional upper limit of normal (ULN).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must be able to understand and sign an Institutional Review Board (IRB) approved informed consent form.
* Patients must have whit blood count (WBC) of 3000 or greater, platelets of 100,000 or greater, and hemoglobin of 9.0 gm/dl or more.
* Patients must be seropositive for Epstein-Barr virus (EBV).
* Patients with unresectable stages III/IV uveal melanoma and metastatic mucosal melanoma will be eligible for this trial.

Exclusion Criteria:

* Patients who are undergoing or have undergone in the past month any other therapy for their melanoma, including radiation therapy, chemotherapy and adjuvant therapy.
* Have major systemic infections, coagulation disorders, or other major medical illnesses (MI) of the cardiovascular or respiratory systems, or have had a documented MI in the last 6 months.
* Require steroid therapy.
* Are pregnant or lactating.
* Are known to be positive for hepatitis BsAg, Hepatitis C or human immunodeficiency virus (HIV) antibody, since cells for DC cannot be grown in the laboratory when virus contaminated.
* Have a prior history of uveitis or autoimmune inflammatory eye disease.
* Have previously received the gp100 209-217 (210M), MART-1 26-35 (27L), gp100 280-288 (288V), tyrosinase 207-215 or NY-ESO-1 157-165 (165V) peptides.
* Have had another malignancy other than cervical carcinoma-in-situ or basal cell

  /squamous cancer of the skin, unless they have undergone curative therapy more than 5 years ago and are still free of detectable disease.
* Since this trial increase the risk of immunological impairment, patients with the following will be excluded from this trial: Hypogammaglobulinemia, Lymphocytopenia, History of impaired immune response, tuberculosis (TB) or positive purified protein derivative (PPD) unless they have received BCG vaccine.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 years, 6 months
  Overall Survival is defined as the time from first day of treatment to time of death due to any cause. If a patient is still alive, survival time is censored at the time of last follow-up.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 3 years, 6 months
  Progression-Free Survival is defined as the time from first day of treatment to the first observation of disease progression or death due to any cause. If a patient has not progressed or died, progression-free survival is censored at the time of last follow-up. Evaluation of target lesions: Progressive Disease (PD)- At least a 20% increase in the sum of longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time to Progression (TTP) | 3 years, 6 months
  Time to Progression is defined as the time from first day of treatment to the first observation of disease progression or death due to disease. If failure has not occurred, failure time is censored at the time of last follow-up. Evaluation of target lesions: Progressive Disease (PD)- At least a 20% increase in the sum of longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States